CLINICAL TRIAL: NCT06446453
Title: Echography-guided Surfactant THERapy (ESTHER) For Preterm Infants With Respiratory Failure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Connecticut Children's Medical Center (Other)
Responsible Party: Principal Investigator, Jacob, Neonatal-Perinatal Fellow, Connecticut Children's Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-005-CCMC
Record Dates: First submitted 2024-06-01; First posted 2024-06-06 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Respiratory Distress Syndrome, Newborn; Pulmonary Surfactants; Intensive Care Units, Neonatal
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): The control group will receive surfactant therapy based on our unit's current surfactant guidelines, including but not limited to a FiO2 requirement ≥ 0.3 on non-invasive positive pressure ventilation.
- Treatment (Experimental): The treatment group will receive surfactant therapy if the initial LUS at 1-2 hours of life is > 9 or if they meet our unit's current surfactant therapy guidelines (irrespective of the LUS).
  Interventions: Diagnostic Test: Echography-guided Surfactant THERapy (ESTHER)

INTERVENTIONS:
Diagnostic Test: Echography-guided Surfactant THERapy (ESTHER) — Decision to administer surfactant therapy using a semi-quantitative lung ultrasound score.
  Arms: Treatment

SUMMARY:
Point-of-care ultrasound (POCUS) is the use of ultrasound by the bedside provider in real time to answer a specific question and guide medical management. POCUS can be used to diagnose the severity of neonatal respiratory distress syndrome (RDS) through a lung ultrasound score. Lung ultrasound scores have also been shown to predict if an infant is treated with an initial dose of surfactant. Therefore, using lung ultrasound scores to guide surfactant therapy for RDS will likely lead to earlier surfactant therapy and may improve short-term respiratory outcomes. This study will test this theory by comparing lung ultrasound score-guided surfactant therapy for premature infants with RDS with our current surfactant administration guidelines.

ELIGIBILITY:
Inclusion Criteria:

* The infant's parent/legal guardian can understand and willingly sign a written informed consent document for this study
* Birth gestational age between 27w0d-36w6d
* Diagnosis of respiratory failure secondary to RDS requiring respiratory support with non-invasive positive pressure ventilation

Exclusion Criteria:

* Unable to obtain lung ultrasound between 1-2 hours of life
* Infants already intubated or received surfactant before the point of care lung ultrasound
* Infants born with congenital cardiac disease, congenital lung disease, or congenital facial/airway malformations
* Infants born with chromosomal abnormalities
* Infants with APGARs ≤ 5 at 10 minutes of life
* Infants requiring cardiopulmonary resuscitation or therapeutic hypothermia in the first 6 hours of life

Ages: 0 Hours to 2 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Estimated)
Dates: Start 2024-06-25 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Oxygen Saturation Index | At 24 hours of life.
  (CPAP Level x FiO2)/(SpO2)

SECONDARY OUTCOMES:
Oxygen Saturation Index | At 48 and 72 hours of life.
  (CPAP Level x FiO2)/(SpO2)

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Kelner, Principal Investigator — Connecticut Children's
Locations (1):
- Connecticut Children's, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No